CLINICAL TRIAL: NCT00883311
Title: A Clinical Usage Study to Evaluate the Safety and Efficacy of BRT-FC-83C in the Management of Mild to Moderate Atopic Dermatitis
Brief Title: A Study of BRT-FC-83C for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomed Research & Technologies, Inc. (Industry)
Responsible Party: Nathan S. Trookman, M.D./Principal Investigator, Thomas J. Stephens & Associates, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRT-C09-C017
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Atopic Dermatitis
Keywords: Efficacy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BRT-FC-83C — BRT-FC-83C is a topical cream to treat atopic dermatitis. It is applied topically, twice a day, to the atopic dermatitis skin lesion for six weeks.

SUMMARY:
The purpose of the study is to determine whether the topical application of BRT-FC-83C is effective in the treatment of mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis is a common skin disease. BRT-FC-83C is a skin cream that does not contain corticosteroids or other anti-inflammatory components. It represents a novel class of skin barrier repair therapy for chronic dermatoses. The objective of this clinical study is to determine whether BRT-FC-83C, applied twice a day to the affected area of the skin, ameliorates signs and symptoms of mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically verified mild to moderate atopic dermatitis. Atopy diagnosis based on clinical scores of 3-7.5 based on the Rajka and Langeland criteria
* Men or women ages 18-50 years
* At least one mild to moderate atopic lesion involving no more than 20% Body Surface Area (BSA)
* Active atopic dermatitis for at least 3 years
* Willingness to cooperate and participate by following study requirements
* Written informed consent

Exclusion Criteria:

* Individuals with actively oozing atopic lesions
* Individuals who are smokers
* Individuals with insulin-dependent diabetes mellitus
* Individuals that are known to be pregnant, nursing, or planning to become pregnant within the next six months after enrollment
* Individuals currently participating in another clinical usage study that would interfere with this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in mean Atopic Dermatitis Severity Index (ADSI) in lesional skin at target site | Eight weeks

SECONDARY OUTCOMES:
Change in mean Trans Epidermal Water Loss (TEWL) in lesional skin at target site | Eight weeks
Change in mean corneometer measurement in lesional skin at target site | Eight weeks
Self assessment of efficacy of BRT-FC-83C on signs and symptoms of atopic dermatitis | Eight weeks
Change in Investigator's Global Assessment (IGA) in lesional skin at target site | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nathan S. Trookman, M.D., Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (1):
- Thomas J. Stephens & Associates, Inc., Colorado Springs, Colorado, United States